CLINICAL TRIAL: NCT03784690
Title: Individualized Blood Pressure Management in Patients Undergoing Cardiac Surgery. A Pilot, Randomized Controlled Study
Brief Title: Individualized Blood Pressure Management in Patients Undergoing Cardiac Surgery
Acronym: PRECISE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: According to new guidelines, the use of vasopressors to force the MAP during CPB at values higher than 80 mmHg is not recommended.
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19
Record Dates: First submitted 2018-10-03; First posted 2018-12-24 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Surgery
Keywords: Hypotension; Intraoperative blood pressure; Cardiopulmonary bypass; Myocardial infarction; Acute kidney injury
MeSH Terms: conditions — Hypotension; Myocardial Infarction; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized BP group (Experimental): Individualized intraoperative BP management
  Interventions: Other: Individualized intraoperative BP management
- Standard treatment group (Placebo Comparator): Standard intraoperative BP management
  Interventions: Other: Standard intraoperative BP management

INTERVENTIONS:
Other: Individualized intraoperative BP management — In the treatment group, the nurse will measure resting blood pressure three times in the ward one day before surgery (after a 5-min rest while lying supine). Average measurement will be used to calculate mean arterial pressure (MAP).
  Before and after CPB patients will receive continuous infusion of norepinephrine to maintain MAP within ± 10% of patients resting MAP. If targeted MAP during CPB could not be achieved after increasing pump-flow (not more than 130%), infusion of norepinephrine will used. After CPB, the choice of vasopressors/inotropes to maintain predefined MAP will be left on attending anesthesiologists based on patient status.
  Arms: Individualized BP group
Other: Standard intraoperative BP management — Standard treatment strategy will be used aiming to maintain pre-bypass and post-bypass MAP at 65-75 mm Hg. MAP during CPB will be maintained at 50-60 mm Hg. If MAP of 50-60 mm Hg during CPB could not be achieved after increasing pump-flow (not more than 130%), infusion of norepinephrine will be started. No vasodilators will be used if MAP will exceed predefined range.
  Arms: Standard treatment group

SUMMARY:
This pilot randomized-controlled study will determine the feasibility of large study comparing individualized versus standard blood pressure (BP) management in patients undergoing cardiac surgery under cardiopulmonary bypass (CPB). Our hypothesis is that maintaining higher BP levels based on preoperative measurements will reduce the incidence of major complications (composite outcome).

DETAILED DESCRIPTION:
Adequate hemodynamic control is a cornerstone in management in patients undergoing different types of surgery. Among all perioperative risk factors, the association between perioperative hypotension and adverse clinical outcomes in noncardiac and cardiac surgery patients is well defined.

Numerous factors are responsible for development of perioperative hypotension. They include but not limited to perioperative use of renin-angiotensin-aldosterone system and calcium channel blockers, hypovolemia, hemodilution, bleeding and inflammatory response syndrome.

To date, several evidence has been accumulated indicating that intraoperational hypertension can be hazardous.

It was shown that even short durations (1 to 5 min) of an intraoperative mean arterial pressure < 55 mmHg were associated with myocardial injuries and acute kidney injury (AKI).

Results of recent large retrospective cohort study conducted in adult patients who underwent cardiac surgery requiring CPB showed that postoperative stroke was strongly associated with sustained mean arterial pressure of less than 64 mmHg during cardiopulmonary bypass.

In patients undergoing CABG the overall incidence of combined cardiac and neurologic complications was significantly lower in the group where MAP during CPB was relatively high (80-110 mmHg) than in the low pressure group (MAP 50-60 mmHg) (p = 0.026). For each of the individual outcomes the trend favored the high pressure group.

Therefore, MAP may be an important intraoperative therapeutic hemodynamic target to reduce the incidence of complications in patients undergoing CPB.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Signed informed consent
* Elective cardiac surgery under CPB (CABG or valve surgery)

Exclusion Criteria:

* Unstable Coronary Artery Disease: Recent (< 6 weeks) myocardial infarction, unstable angina, severe (> 70%) left main coronary artery stenosis
* Uncontrolled hypertension preoperatively (SBP > 160 mm Hg)
* Critical preoperative state (ventricular tachycardia or ventricular fibrillation or aborted sudden death, preoperative cardiac massage, preoperative ventilation before anesthetic room, hemodynamic instability, preoperative inotropes or intraaortic balloon pumping, preoperative severe acute renal failure (anuria or oliguria <10ml/hr)
* Planned surgery on aorta
* Emergency surgery
* Pregnancy
* Current enrollment into another randomized controlled trial (in the last 30 days)
* Previous enrollment and randomization into current study
* Glomerular filtration rate ≤59 ml/min/1.73m2 (Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
Compliance with the protocol | Operative day 1
  Successful compliance with protocol is defined as ≥ 90% of prescribed intervention being administered across all patients.
Successful recruitment rate | 12 month
  Successful recruitment rate will be defined as recruitment of 2 patients per week.

SECONDARY OUTCOMES:
Postoperative creatinine concentration | 3 days after surgery
  Plasma creatinine level will be measured daily during 3 postoperative days.
Postoperative cardiac troponin I level | 12 hours after surgery
  Cardiac troponin I level wil be measured in the time frame from 6 to 12 hours postoperatively.
Intraoperative blood pressure | Operative day 1
  Intraoperative blood pressure (mean, systolic and diastolic) will be registered every 5 minutes intraoperatively using invasive blood pressure monitoring system.
Rate of postoperative complications | 30 days after surgery
  Postoperative complications (myocardial infarction, atrial fibrillation, stroke, delirium, need for renal replacement therapy, infection, reexploration for bleeding) will be defined according to standard European Society of Anaesthesiology/European Society of Intensive Care Medicine definitions where possible.
Postoperative blood loss | Postoperative day 1
  Drainage volume (ml/kg) will be measured in the next morning after surgery.
Daily Sequential Organ Failure Assessment (SOFA) score | 30 days after surgery
  Organ failure will be assessed by using Sequential Organ Failure Assessment (SOFA) score which will be recorded daily until patient discharge from the ICU. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The score ranges from 0 to 24 points (the higher the score, the higher the mortality).
Peak concentration of lactate during CPB and up to 24 hours after surgery | Postoperative day 1
  Lactate values (mmol/l) will be measured every 6 hours during the first 24 postoperative hours.
Oxygen delivery during CPB | Operative day 1
  Oxygen delivery during CPB will be calculated according to the standard formula (pump flow x O2 arterial content).
Cerebral oxygenation (near infrared spectroscopy) | Operative day1
  Number of cerebral desaturations will be recorded intraoperatively.
Ventilation > 24 hours | 30 days after surgery
  Number of patients with duration of ventilation more than 24 h.
Duration of ICU stay and hospitalization | 30 days after surgery
  Number of postoperative days spent in the ICU and in the hospital will be counted.
30-day all-cause mortality | 30 days after surgery
  Number of patients who will die within 30-day after surgery from any cause
Need for blood transfusions | 30 days after surgery
  Number of patients who will need transfusions of any blood products (RBC, fresh frozen plasma, platelets, cryoprecipitate).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lomivorotov, MD, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI, Khanna AK. Perioperative myocardial injury and the contribution of hypotension. Intensive Care Med. 2018 Jun;44(6):811-822. doi: 10.1007/s00134-018-5224-7. Epub 2018 Jun 4. PMID 29868971
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Gold JP, Charlson ME, Williams-Russo P, Szatrowski TP, Peterson JC, Pirraglia PA, Hartman GS, Yao FS, Hollenberg JP, Barbut D, et al. Improvement of outcomes after coronary artery bypass. A randomized trial comparing intraoperative high versus low mean arterial pressure. J Thorac Cardiovasc Surg. 1995 Nov;110(5):1302-11; discussion 1311-4. doi: 10.1016/S0022-5223(95)70053-6. PMID 7475182